CLINICAL TRIAL: NCT03753321
Title: Comparison of the Effect of Whey and Soy Protein Supplementation on Muscle Damage Markers and Performance After a Speed Endurance Training Protocol in Football Players
Brief Title: Whey and Soy Protein Supplementation in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: WHEY vs SOY PROTEIN - UTH
Record Dates: First submitted 2018-10-12; First posted 2018-11-26 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Skeletal Muscle Damage; Muscle Damage; Athletic Performance
MeSH Terms: interventions — Whey Proteins; Soybean Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey protein (Experimental): Whey protein isolate supplementation (7 day pre-loading phase and 3 day training phase). The protein dose will be individually adjusted to reach a total protein intake of 1.5 g protein/kg body mass/day.
  Interventions: Dietary Supplement: Whey protein
- Soy protein (Experimental): Soy protein isolate supplementation (7 day pre-loading phase and 3 day training phase). The protein dose will be individually adjusted to reach a total protein intake of 1.5 g protein/kg body mass/day.
  Interventions: Dietary Supplement: Soy protein
- Placebo (maltodextrin) (Placebo Comparator): Isoenergetic, maltodextrin (7 day pre-loading phase and 3 day training phase)
  Interventions: Dietary Supplement: Placebo (maltodextrin)

INTERVENTIONS:
Dietary Supplement: Whey protein — Whey protein isolate supplementation, individually adjusted to reach a total protein intake of 1.5 g/kg body weight/day for 10 days (7 days pre-loading and 3 days during trials 1 and 2)
  Arms: Whey protein
Dietary Supplement: Soy protein — Soy protein isolate supplementation, individually adjusted to reach a total protein intake of 1.5 g/kg body weight/day for 10 days (7 days pre-loading and 3 days during trials 1 and 2)
  Arms: Soy protein
Dietary Supplement: Placebo (maltodextrin) — Isoenergetic placebo (maltodextrin) for 10 days (7 days pre-loading and 3 days during trials 1 and 2
  Arms: Placebo (maltodextrin)

SUMMARY:
In a constant effort to find ways to make a quicker recovery between demanding workouts and football matches, this study is the first to investigate the benefits of protein supplementation, and compares two types of proteins, an animal-derived (whey) and a plant-derived (soy) protein, after an exercise-induced muscle injury caused by a speed endurance training protocol. Soy protein could be a cheaper and more environment-friendly alternative for athletes involved in high-velocity strength training.

DETAILED DESCRIPTION:
A randomized, three-trial (placebo vs. whey protein isolate vs. soy protein isolate consumption), cross-over, double-blind design.

1. Baseline performance testing: Initially, volunteers will participate in a performance testing procedure at University facilities. These measurements include:

   A) measurement of descriptor variables: a) body composition (DXA), b) VO2max, c) Yo-Yo intermittent endurance level 2 (Yo-Yo IE2), d) Yo-Yo intermittent recovery test level 2 (Yo-Yo IR2), e) technical skill level, f) daily dietary intake profile (over a 7-day period), g) gabitual physical activity level (over a 7-day period) and h) resting mtabolic rate (RMR).

   B) Measurement of dependent variables: a) isokinetic strength (concentric, eccentric) and maximal voluntary isometric contraction (MVIC) of knee extensors and flexors of both lower limbs, b) counter movement jump height (CMJ), c) repeated sprint ability (RSA), d) speed (10 and 30 m), e) delayed onset of muscle soreness (DOMS), f) blood sampling for measurement of lactate concentration, creatine kinase activity (CK) and inflammatory markers [i.e.Glutathione (GSH), total antioxidant capacity (TAC) and protein carbonyls (PC)].
2. A 1-week adaptive period: based on a dietary analysis, participants will be given a dietary plan [taking into account the resting metabolic rate (RMR) and total daily physical activity related energy expenditure], providing a standard protein intake of 0.8-1 g protein/kg/day over the 1-week adaptive period. This protein intake is accepted as the average and population-safe protein intake during periods of very low physical activity and/or exercise levels. RMR, daily dietary intake and physical activity will be measured before the adaptive period. Familiarization with the training protocol will take place during this phase.
3. Participants will randomly participate in three trials including: whey protein (WP), soy protein (SP) and placebo (PL) supplementation:

   * A 7-day pre-loading phase: A 7-day pre-loading phase will be applied prior to each trial, during which volunteers will receive the respective supplement (placebo, whey protein or soy protein). In WP and SP trials, participants will consume daily the appropriate amount of protein to reach a total protein intake of 1.5 g protein/kg body weight (BW).
   * On the 7th day (end of pre-loading phase), participants will repeat performance testing (assessment of all dependent variables according to baseline testing) and blood sampling.
   * On the 8th day, participants will perform the speed-endurance production training (SEPT) session 1 (1st trial). During training, participants internal (heart rate) and external load (total distance, speed zones, acceleration and decelerations, impacts) will be continuously monitored using heart rate monitors and global positioning system (GPS) instrumentation.
   * Immediately after the training protocol: Determination of blood lactate concentration (3-4 minutes post-training) and assessment of MVIC (1 hour, 2 hours and 3 hours post-training).
   * 1-Day post-training (9th day; 24 hours post-training): Blood sampling (for the determination of CK, GSH, TAC and PC) and measurement of dependent variables (i.e. isokinetic strength, MVIC, Speed, RSA, CMJ and DOMS).
   * 2-Days post-training (10th day; 48 hours post-training): Blood sampling (for the determination of CK, GSH, TAC and PC) and assessment of DOMS. Thereafter, the SEPT session 2 will take place during which the particpants' internal and external load will be continuously monitored (as described in SEPT session 1).
4. Wash-out period: 2-week without any activity or supplementation.
5. 2nd trial: repeat of stages 3 and 4.
6. 3rd trial: repeat of stage 3.

ELIGIBILITY:
Inclusion Criteria:

* Playing at a competitive level (top three divisions) for ≥3 years
* Free of any recent history of illnesses, musculoskeletal problems and metabolic diseases
* No use of supplements and medications (for ≤6 months prior to the study)
* Non-smokers

Exclusion Criteria:

* A known milk intolerance or allergy
* A recent febrile illness
* History of muscle lesion
* Lower limb trauma
* Metabolic diseases.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Change in field activity during the speed-endurance production training (SEPT) | Throughout the SEPT sessions in all trials
  Field activity will be continuously recorded during both SEPT sessions using global positioning system (GPS) technology
Change in heart rate during the speed-endurance production training (SEPT) | Throughout the SEPT sessions in all trials
  Heart rate will be continuously recorded during both SEPT sessions using heart rate monitors.
Change in creatine kinase in plasma | Baseline; Post-loading (Day 7); 24 hours (Day 9) and 48 hours (Day 10) following SEPT session 1.
  Concentration of creatine kinase will be measured in plasma
Change in repeated sprint ability (RSA) | Baseline; Post-loading (Day 7); 24 hours (Day 9) following SEPT session 1
  5 x 30 m sprints will be performed with 25 seconds rest in-between
Change in countermovement jump (jump height in centimeters) | Baseline; Post-loading (Day 7); 24 hours (Day 9) following SEPT session 1
  Countermovement jump will be assessed on a contact platform
Change in isokinetic strength of lower limbs | Baseline; Post-loading (Day 7); 24 hours (Day 9) following SEPT session 1
  Isokinetic strength will be assessed on an isokinetic dynamometer for both knee extensors and knee flexors at 60 degrees.
Change in maximal voluntary isometric contraction (MVIC) of lower limbs | Baseline; Post-loading (Day 7); 1, 2 and 3 hours post-SEPT session 1; 24 hours (Day 9) and 48 hours (Day 10) following SEPT session 1.
  MVIC will be assessed on an isokinetic dynamometer for knee extensors at 90 degrees and knee flexors at 30 degrees
Change in delayed onset of muscle soreness | Baseline; Post-loading (Day 7); 24 hours (Day 9) and 48 hours (Day 10) following SEPT session 1.
  Muscle soreness will assessed during palpation of the muscle belly and the distal region of relaxed vastus medialis, vastus lateralis and rectus femoris following three repetitions of of a full squat. Subjects will rate their DOMS on a visual analogue scale (0-10). A score of O indicates no sign or symptom of DOMS, a score of 10 indicated severe signs and symptoms of delayed onset muscle soreness (DOMS). These signs and symptoms include dull, diffuse pain and tenderness; stiffness; swelling; and decreased strength of the exercised muscle.
Change in total antioxidant capacity in plasma | Baseline; Post-loading (Day 7); 24 hours (Day 9) and 48 hours (Day 10) following SEPT session 1.
  Total antioxidant capacity will be measured in plasma
Change in protein carbonyl levels in plasma | Baseline; Post-loading (Day 7); 24 hours (Day 9) and 48 hours (Day 10) following SEPT session 1.
  Protein carbonyl levels will be measured in plasma
Change in GSH levels in red blood cell lysate | Baseline; Post-loading (Day 7); 24 hours (Day 9) and 48 hours (Day 10) following SEPT session 1.
  GSH will be measured in red blood cell lysate
Change in sprint time | Baseline; Post-loading (Day 7); 24 hours (Day 9) following SEPT session 1
  Sprint time will be assessed over a 10m and 30m distance using light cells.

SECONDARY OUTCOMES:
Dietary intake | Over a 7-day period at baseline.
  Dietary intake will be assessed using 7-day diet recalls.
Concentration of blood lactate | Pre- and Post-SEPT session 1 (Day 8), Pre- and Post-SEPT session 2 (Day 10)
  Blood lactate will be measured using an automatic analyzer
Change in habitual physical activity | Over a 7-day period at baseline
  Physical activity will be measured using 3-axial accelerometers
Change in resting metabolic rate (RMR) | At baseline.
  RMR will be measured using open-circuit indirect calorimeter with a ventilated hood system, after an overnight fast.
Change in body composition | At baseline.
  Body composition will be assessed using dual-energy X-ray absorptiometry (DXA).
Change in maximal oxygen uptake | At baseline.
  Maximal oxygen uptake (VO2max) will be measured during a graded exercise testing on a treadmill, by using open-circuit spirometry with an automated online pulmonary gas exchange system, via breath-by-breath analysis.
Change in soccer-specific conditioning. | At baseline.
  Soccer-specific conditioning will be assessed using the the Yo-Yo intermittent endurance level 2 test (Yo-Yo IE2) and the Yo-Yo intermittent recovery level 2 test (Yo-Yo IR2).

CONTACTS AND LOCATIONS:
Overall Officials: Savvas Kritikos, MScc, Principal Investigator — UNIVERSITY OF THESSALY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES
Locations (1):
- Exercise Biochemistry Laboratory, School of Physical Education & Sports Sciences, University of Thessaly, Trikala, Greece

REFERENCES:
- [Derived] Kritikos S, Papanikolaou K, Draganidis D, Poulios A, Georgakouli K, Tsimeas P, Tzatzakis T, Batsilas D, Batrakoulis A, Deli CK, Chatzinikolaou A, Mohr M, Jamurtas AZ, Fatouros IG. Effect of whey vs. soy protein supplementation on recovery kinetics following speed endurance training in competitive male soccer players: a randomized controlled trial. J Int Soc Sports Nutr. 2021 Mar 16;18(1):23. doi: 10.1186/s12970-021-00420-w. PMID 33726784